CLINICAL TRIAL: NCT03030456
Title: Evaluation of the Effects of Whole Body Vibration Training on Functional Capacity, Muscle Strength, and Biochemical Profile in Elderly Women
Brief Title: Whole Body Vibrations on Functional Capacity, Muscular Strength, and Biochemical Profile in Elders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Santa Cruz do Sul (Other)
Responsible Party: Principal Investigator, Greice Raquel Machado, PHYSICAL THERAPIST, University of Santa Cruz do Sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 57756916.0.0000.5343
Record Dates: First submitted 2016-09-21; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Aging; Oxidative Stress
Keywords: whole body vibration; Oxidative Stress; Aged; Biochemical profile; muscle strength; flexibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Elderly women receiving a list of general health orientations through an 8 week period
- Power Plate® (Experimental): Power Plate®: training of elderly women
  Interventions: Device: Power Plate®

INTERVENTIONS:
Device: Power Plate® — Training of elderly women with Whole Body Vibrations through the use of a vibratory platform.
  Other Names: Whole Body Vibrations
  Arms: Power Plate®

SUMMARY:
This study is a randomized clinical trial that has as objective to evaluate the effects of training with a vibratory platform on body composition, muscular strength functional capacity, flexibility and biochemical profile on elderly women. It will be done in the city of Santa Cruz do Sul, Rio Grande do Sul, with elderly women between the ages of 60 and 80 years-old, within the municipal limits and nearby areas selected randomly by a brown envelope in which a note will be stating if they belong to the control or vibratory platform group, in which the participant will be receiving whole body vibrations on the platform. The recruiting will be done by the institution through e-mail or by public call.

Women will be evaluated through anamesis. On the evaluation, a questionaire will be applied, in order to evaluate if they don´t have counterindications for the vibratory platform. They will be evaluated in their general health, socio-economical status, and history of physical activity. Participants will have their doubts cleared about the study, and a written consent will be signed. Before the intervention with whole body vibrations, nutritional and physical activity aspects will be evaluated. The treatment period on the vibratory platform will be of 8 weeks, before and after it, anthropometrical, biochemical, strength, flexibility, palmar prehension strength, metabolic basal load, and functional capacity measurements will be taken. Before and after every session on the vibratory platform, heart rate, respiratory rate, arterial pressure, and peripheric oxygen saturation will be evaluated. The interventional procedure will be done with a vibratory platform (Power Plate®, model my7™, UK) with a frequency of 30 - 40 Hz, with low (2mm) or high (4mm) amplitude. Training will last 8 weeks with 3 sessions per week, lasting between 30 seconds and 1 minute of training, and 30 seconds to 1 minute of rest, with the subject positioned in orthosis with a knee flexion of 15° and a feet width distance of 20 cm. The frequency will be of 35 Hz and the amplitude of 2 mm.

The study aims to contribute with reducing the body mass index and body fat percentage, to improve the lean mass, palmar prehension strength, muscular strength on the lower limbs and flexibility, also obtaining better biochemical profiles after the training period.

DETAILED DESCRIPTION:
After evaluating the anamnesis and having the written consent signed and clarified, the elderly women will be evaluated before and after the intervention period of 8 weeks of training on the vibratory platform. First, academics from the nutrition degree of the University of Santa Cruz do Sul (UNISC) will perform nutritional evaluations on the subjects, asking them their 24 hour eating habits, there will not be any interference on the subjects diet, also they will have to keep these habits until the end of the trial. Then there will be a socio-economical indicators evaluation through a questionnaire of socio-economical classification from the Brazilian Association of Research Companies.The evaluation of their level of physical activity will be done by the International Physical Activity Questionnaire. The anthropometrical evaluation will consider height, weight, body mass index, waist circumference, hip circumference, and hip-waist ratio. Body fat percentage, lean mass, and basal metabolic rate will be obtained through bioimpedance (Biodynamics 450, USA), recommending 5 hours fasting prior to the procedure. Biochemical tests will be done collecting blood at the University of Santa Cruz Exercise Biochemistry Laboratory, on the following variables: hemogram, glycemia, cholesterol, triglycerides, Urea, creatine, uric acid. Oxidative stress evaluation with the Thiobarbituric acid reactive substances (TBARS) test will be done after urine collection once a week, before intervention and immediately after the session. Control group subjects will have urine collected twice: on the day when cards will be handed in and on the last day of evaluations. Physical evaluation will be done in the week prior to the intervention with the vibratory platform and in the last week of treatment, where flexibility through Wells Bank will be evaluated, as well as lower limb muscular strength by the maximum repetitions test, and palmar prehension strength will be obtained through dynamometer. Functional Capacity will be evaluated with the six minute walk test.

The intervention procedure with the vibratory platform (Power Plate®, model my7™, UK) will last 8 weeks, 3 times a week with work periods lasting between 30 seconds and 1 hour and rest periods of 30 seconds to 1 minute with a total session time of 10 to 20 minutes. The individual will be then positioned in orthosis with a knee flexion of a 15° and a foot width distance of 20 cm. A frequency of 35 Hz and an amplitude of 2 mm will be used. The protocol with number of session, time of session, time of vibrations and rest, is as follows: 1st through 6th session, total time of 10 minutes, with 30 seconds of vibration alternated with 1 minute rest; 7th through 12th session, total time of 10 minutes, vibrations and rest time of 1 minute each; 13th trough 18th session, total session time of 15 minutes, vibrations and rest time of 1 minute each, 19th through 24th session, total time of 20 minutes, time of vibration 1 minute and rest time of 30 seconds.

Statistical analysis: This will be done using the Statistical Package for Social Science (Version 23.0 USA) program. To test data normality the investigators will use the Kolmogorov-Smirnov test. Parametric data will be presented in mean and standard deviation and non-parametric data in median and interquartile intervals. The intragroup deltas from the pre and post training periods on the vibratory platform on both groups will be evaluated through Student´s T Test (paired T test or non-parametric equivalent for intergroup comparisons).

To evaluate body composition, metabolic rate, palmar prehension strength, flexibility, muscular strength, distance traveled through the Six minute walking test (6SMWT), biochemical profile and oxidative stress between the groups evaluated pre and post training period, a Student´s T test will be used. Significance level will be p < 0,05.

Sample size: It was based on a previous study by Rees et al. (2008). To detect a difference of 8,9 W/Kg between knee flexion torque pre and post training on the vibratory platform, considering a p value < 0,05, a statistical power of 80% and a 10% loss, 34 subjects will be needed in each group to be evaluated in pre and post training.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 60 or older.
* Non-physical activity practicing elderly women.
* Maximum weight of 159 kg.
* BMI between 18 and 39 kg/m².

Exclusion Criteria:

* Systemic arterial hypertension, (systolic arterial pressure >140 mmHg or diastolic arterial pressure >90 mmHg).
* Cognitive compromising neutropenia.
* Individual subject to surgical procedures, where bone prosthetics has been implanted or cardiac pacemaker.
* Individuals diagnosed with labyrinthitis, disc hernia, thrombosis,decompensated diabetes or cancer.
* Cognitive deficit.
* Orthopedic deficit which makes participation impossible.
* Persistent discomfort after using the vibratory platform.
* Individuals missing three consecutive training sessions on the vibratory platform.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-01 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Effects of whole body vibrations training on Functional Capacity in Elderly Women. | eight weeks
  Functional Capacity will be measured through distance traveled with the six minute walk test.
Effects of whole body vibrations training on Muscle Strength in Elderly Women. | eight weeks
  Muscular strength will be measured by the maximum repetitions test.
Effects of whole body vibrations training on Biochemical Profile in Elderly Women. | eight weeks
  Biochemical profile will be measured through blood collection and there will be a result (number) for each one of the following variables: hemogram, glycemia, cholesterol, triglycerides, Urea, creatine, uric acid. Oxidative stress will be measured through TBARS test, which will present a numerical result.

CONTACTS AND LOCATIONS:
Overall Officials: Greice Raquel Machado, Principal Investigator — Masters Student

IPD SHARING:
Plan to Share IPD: No